CLINICAL TRIAL: NCT05068011
Title: Differential Target Multiplexed Spinal Cord Stimulation: a Multicenter Cohort Study
Brief Title: Differential Target Multiplexed Spinal Cord Stimulation
Acronym: DETECT
Status: Recruiting | Type: Observational
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: DETECT
Record Dates: First submitted 2021-09-09; First posted 2021-10-05 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Failed Back Surgery Syndrome; Persistent Spinal Pain Syndrome Type 2
Keywords: differential target multiplexed spinal cord stimulation
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal cord stimulation: Patients will receive differential target multiplexed spinal cord stimulation
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — differential target multiplexed stimulation

SUMMARY:
Evaluation of the effectiveness of differential target multiplexed spinal cord stimulation for treatment of chronic back and leg pain. Additionally, a subgroup analysis will be performed to evaluate potential differences between paddle/surgical leads versus percutaneous leads.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe chronic pain (> 5 on numeric rating scale, NRS) for at least 6 months due to FBSS (PSPS T2) and suitable for treatment with DTM SCS according to the treating physician
* Age > 18 years
* Patient has been informed of the study procedures and has given written informed consent
* Patient willing to comply with study protocol including attending the study visits

Exclusion Criteria:

* Expected inability of the patient to receive or properly operate the spinal cord stimulation system
* History of coagulation disorder, lupus erythematosus, diabetic neuropathy, rheumatoid arthritis, or morbus Bechterew
* Active malignancy
* Addiction to drugs, alcohol (>5 units per day) and/or medication
* Evidence of an active disruptive psychiatric disorder or other known condition that may impact perception of pain, compliance to the intervention, and/or ability to evaluate treatment outcome as determined by investigator
* Immune deficiency (e.g. HIV positive, immunosuppressive treatment)
* Life expectancy < 1 year
* Local infection or any other skin disorder at site of incision
* Pregnancy
* Other implanted active medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic back and leg pain due to Failed Back Surgery Syndrome (FBSS)/Persistent Spinal Pain Syndrome type 2 (PSPS-T2), who will receive treatment with differential target multiplexed (DTM) SCS.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall pain intensity with Visual Analogue Scale (VAS) | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Overall pain, defined as a combination of back and leg pain, but not pain from other body parts, measured with the VAS (100mm)

SECONDARY OUTCOMES:
Back pain intensity with Visual Analogue Scale (VAS) | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
Leg pain intensity with Visual Analogue Scale (VAS) | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
Pain medication use | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Open question regarding the dosage, frequency and type of pain medication
Functional disability | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The functional disabilities will be assessed with the Oswestry Disability Index (ODI)
Health related quality of life | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Health related quality of life, evaluated with the EuroQol with five dimensions and 5 levels
Patient global impression of change | Evaluated at 1 month, 6 months and 12 months of DTM SCS.
  Patients will be asked to quantify the impression of change after treatment using the Patient Global Impression of Change scale (PGIC).
Clinical holistic responder status | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
Patients' individual competencies for self-management | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Patient activation measure-13 (PAM) is a 13-item instrument which assesses self-reported behaviour, knowledge, and confidence for self-management of one's health.
Work status | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Work status is evaluated with a self-designed questionnaire
Pain catastrophizing | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The Pain Catastrophizing Scale (PCS) will be used to measure the level of pain catastrophizing
Symptoms of central sensitisation. | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The Central Sensitization Inventory is used to measure symptoms of central sensitisation
Anxiety and Depression. | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The hospital Anxiety and Depression Scale (HADS) will measure symptoms of anxiety and depression
Healthcare utilisation. | The change between implantation and evaluation at 1 month, 6 months and 12 months of DTM SCS
  Postoperative healthcare expenditure will be investigated by self-reporting methods.
Time spent in body postures | The data will be extracted from SCS implantation up to 1 month of SCS, from 1 month of SCS up to 6 months and from 6 months up to 12 months
  Based on the AdaptiveStim technology, the time spent in body postures can be recorded.
(Serious) adverse events | Throughout study period
  Systematically recording all adverse events
Proportion of successful DTM trials. | Evaluated after final SCS implantation
Battery consumption | Registration at 1 month, 6 months and 12 months of DTM SCS
Prevalence of technical issues with regard to DTM SCS programming | Throughout study period
DTM SCS stimulation parameters | Registration at 1 month, 6 months and 12 months of DTM SCS
Patient expectations concerning SCS | Evaluated at baseline visit
  Self-constructed open question to evaluate patient expectations about SCS

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (14):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - ZNA, Antwerp
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - AZ Sint-Lucas Brugge, Bruges
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - Heilig Hart Ziekenhuis Lier, Lier
  - Centre Hospitalier Régional (CHR) de la Citadelle, Liège
  - AZ Sint-Maarten, Mechelen
  - AZ Delta, Roeselare
  - Vitaz, Sint-Niklaas
  - AZ Turnhout, Turnhout
  - GZA, Wilrijk

REFERENCES:
- [Derived] Goudman L, De Smedt A, Eldabe S, Rigoard P, Billot M, Roulaud M; DETECT consortium; Moens M. Differential target multiplexed spinal cord stimulation in patients with Persistent Spinal Pain Syndrome Type II: a study protocol for a 12-month multicentre cohort study (DETECT). BMJ Open. 2024 Nov 9;14(11):e083610. doi: 10.1136/bmjopen-2023-083610. PMID 39521475